CLINICAL TRIAL: NCT03155412
Title: Limited Adipose Tissue Expandability as a Risk Factor for Development of Type 2 Diabetes: the Role of Preadipocytes
Brief Title: Adipose Tissue Expandability and Type 2 Diabetes
Acronym: LIMEX
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Vladimir Stich, Professor, MUDr, Charles University, Czech Republic
Other Study IDs: 16-14048S
Record Dates: First submitted 2017-05-15; First posted 2017-05-16 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Type2 Diabetes Mellitus
Keywords: Type 2 Diabetes; adipose tissue; preadipocytes; expandability; hypertrophy; hyperplasia; lipogenesis; adipogenesis; insulin sensitivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertrophy; Hyperplasia; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — adipose tissue plasma / serum preadipocytes (cells)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Offspring of type 2 diabetic patients: Group 1: 25 healthy lean men (age 30-45, BMI <28) with genetic predisposition for type 2 diabetes mellitus (T2DM) - i.e. their two first-degree relatives (parents, siblings) or one first-degree relative and two second-degree relatives with type 2 diabetes (grandparents, uncle, aunt) were diagnosed with T2DM. Exclusion criteria: any prior history of obesity, elevated triglyceride concentration, hypertension, thyroid or other endocrine disease, smoking, drug abuse.
- Control subjects: Group 2: 25 healthy lean men (age 30-45, BMI <28) without any family history of T2DM. Exclusion criteria: any prior history of obesity, elevated triglyceride concentration, hypertension, thyroid or other endocrine disease, smoking, drug abuse. Subjects matched for BMI, fat mass and age to subjects in Group 1 will be recruited.

SUMMARY:
The goal of the study is to analyze deviations in adipogenic potential and metabolic properties of preadipocytes in subjects with genetic predisposition to type 2 diabetes, and thus identify factors that underlie hypertrophic growth of adipose tissue associated with the development of this disease.

DETAILED DESCRIPTION:
Adipose tissue (AT) expands in response to excessive energy intake by hyperplasia or hypertrophy. While hyperplasia is associated with preservation of insulin sensitivity, hypertrophic AT exerts a number of metabolic defects. The mechanisms by which hyperplasia is suppressed at the expense of AT hypertrophy remain unknown, but it is expected that the hypertrophy of adipocytes is primarily driven by insufficient recruitment and differentiation of available preadipocytes. The limitation of hyperplasia occurs already in non-obese healthy subjects who are genetically predisposed to Type 2 Diabetes. Using these and control subjects, the LIMEX project aims to analyze the mechanisms of AT expandability. The project will combine in vivo characterization of AT and in vitro studies on human preadipocytes derived from AT biopsies obtained during clinical study. In vitro, proliferation, adipogenesis and lipogenesis of adipose cells will be monitored and these properties will be related to the degree of AT hypertrophy in vivo, insulin sensitivity and genetic predisposition to metabolic complications.

ELIGIBILITY:
Inclusion Criteria:

* healthy non-obese men
* subject has genetic predisposition for T2DM- i.e. two first-degree relatives (parents, siblings) or one first-degree relative and two second-degree relatives with type 2 diabetes (grandparents, uncle, aunt) diagnosed with T2DM OR
* subject without any family history of T2DM.

Exclusion Criteria:

* any prior history of obesity
* elevated triglyceride concentration (above 1.7 mmol/l)
* hypertension
* thyroid or other endocrine disease
* smoking
* drug abuse

Ages: 30 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 50 healthy lean men (age 30-45, BMI <26). Two groups of subjects (n=25) matched for BMI, fat mass and age.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2016-01; Primary Completion 2018-03 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Adipogenic capacity of preadipocytes | 3 months from the establishment of the cell culture
  proliferation assays, messenger ribonucleic acid (mRNA) gene expression

SECONDARY OUTCOMES:
Insulin sensitivity | 3 hours investigation of the subject at the start of the study
  Glucose disposal measured by hyperinsulinemic-euglycemic clamp
Glucose tolerance | 2 hours investigation of the subject at the start of the study
  Oral glucose tolerance test (OGTT)
Lipid metabolism | 3 months from the establishment of the cell culture
  Lipolysis, lipogenesis in cell cultures of adipocytes derived from the subjects

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Stich, prof, Principal Investigator — Third faculty of medicine, Charles University in Prague
Locations (1):
- Third Faculty of Medicine, Charles University, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guilherme A, Virbasius JV, Puri V, Czech MP. Adipocyte dysfunctions linking obesity to insulin resistance and type 2 diabetes. Nat Rev Mol Cell Biol. 2008 May;9(5):367-77. doi: 10.1038/nrm2391. PMID 18401346
- [Background] Lu Q, Li M, Zou Y, Cao T. Induction of adipocyte hyperplasia in subcutaneous fat depot alleviated type 2 diabetes symptoms in obese mice. Obesity (Silver Spring). 2014 Jul;22(7):1623-31. doi: 10.1002/oby.20705. Epub 2014 Feb 11. PMID 24435986
- [Background] Alligier M, Gabert L, Meugnier E, Lambert-Porcheron S, Chanseaume E, Pilleul F, Debard C, Sauvinet V, Morio B, Vidal-Puig A, Vidal H, Laville M. Visceral fat accumulation during lipid overfeeding is related to subcutaneous adipose tissue characteristics in healthy men. J Clin Endocrinol Metab. 2013 Feb;98(2):802-10. doi: 10.1210/jc.2012-3289. Epub 2013 Jan 2. PMID 23284008
- [Background] Medina-Gomez G, Gray SL, Yetukuri L, Shimomura K, Virtue S, Campbell M, Curtis RK, Jimenez-Linan M, Blount M, Yeo GS, Lopez M, Seppanen-Laakso T, Ashcroft FM, Oresic M, Vidal-Puig A. PPAR gamma 2 prevents lipotoxicity by controlling adipose tissue expandability and peripheral lipid metabolism. PLoS Genet. 2007 Apr 27;3(4):e64. doi: 10.1371/journal.pgen.0030064. PMID 17465682
- [Background] Rossmeislova L, Malisova L, Kracmerova J, Tencerova M, Kovacova Z, Koc M, Siklova-Vitkova M, Viquerie N, Langin D, Stich V. Weight loss improves the adipogenic capacity of human preadipocytes and modulates their secretory profile. Diabetes. 2013 Jun;62(6):1990-5. doi: 10.2337/db12-0986. Epub 2013 Feb 1. PMID 23378611
- [Derived] Koc M, Siklova M, Sramkova V, Stepan M, Krauzova E, Stich V, Rossmeislova L. Signs of Deregulated Gene Expression Are Present in Both CD14+ and CD14- PBMC From Non-Obese Men With Family History of T2DM. Front Endocrinol (Lausanne). 2021 Feb 15;11:582732. doi: 10.3389/fendo.2020.582732. eCollection 2020. PMID 33658980